CLINICAL TRIAL: NCT05925179
Title: Effects of Pre-operative Antibiotics on the Wound Healing Following Clinical Crown Lengthening Surgery
Brief Title: Effects of Antibiotic Prophylaxis on the Healing Parameters Following Surgical Crown Lengthening
Acronym: SCLABP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Mustafa YILMAZ, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Antibiotics crown lengthening
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Tooth Diseases; Tooth Wear
MeSH Terms: conditions — Tooth Diseases; Tooth Wear | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antibiotic prophylaxis (Experimental): per os 2 g augmentin one hour prior to surgery
  Interventions: Procedure: Surgical crown lengthening; Drug: Augmentin
- placebo control (Placebo Comparator): per os placebo one hour prior to surgery
  Interventions: Procedure: Surgical crown lengthening

INTERVENTIONS:
Procedure: Surgical crown lengthening — Surgical clinical crown lengthening with bone excision
Drug: Augmentin — Pre-operative antibiotic prophylaxis (2 g Augmentin)
  Arms: antibiotic prophylaxis

SUMMARY:
The goal of this clinical trial is to test the effects of prophylactic antibiotics in healthy individuals who are in need of surgical crown lengthening. The main question it aims to answer is if single dose antibiotics prior to surgical crown lengthening has any effects on the healing outcomes.

Participants will be asked to take either

* 2 g of amoxicillin + clavulanate, or
* placebo, one hour prior to surgery and without knowing what medicine they took.

Researchers will compare the wound healing and self-reported outcomes of the antibiotics group and placebo group.

ELIGIBILITY:
Inclusion Criteria:

* in need of surgical crown lengthening operation in one/two teeth

Exclusion Criteria:

* systemic diseases which may affect periodontal tissues and/or healing process such as diabetes mellitus
* antibiotic or anti-inflammatory drug use in the last 3 months
* pregnancy/lactation
* chronic steroid, immunosuppressant or NSAD use
* age <18 years
* positive bleeding on probing at the surgical site and/or active periodontal disease
* <2 mm keratinized mucosa at the surgical site following surgery (estimated surgical outcome before the operation)
* Miller 2 or 3 tooth mobility
* penicillin allergy
* unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Early healing index (inflammation phase) | at 3 days
  Scores are given as specified below (Hamzani et al. 2018)
  Bleeding (spontaneous or provoked) Yes: 0; No: 1
  Granulation tissue Yes: 0; No: 1
  Hematoma Yes: 0; No: 1
  Tissue color Redder or whiter than opposite site: 0; Similar to opposite site: 1
  Incision margins Incomplete flap closure/fibrin clot/partial or complete necrosis: 0; Complete closure/fine fibrin line: 1
  Suppuration Yes: 0; No: 1
  Edema VAS 6-10: 0; VAS 1-5: 1
  Pain VAS 6-10: 0; VAS 1-5: 1
Early healing index (proliferation phase) | at 10 days
  Scores are given as specified below (Hamzani et al. 2018)
  Re-epithelization Partial: 0; Complete: 1
  Tissue color Redder or whiter than opposite site: 0; Similar to opposite site: 1
  Scar wider than 2 mm/contour irregularity: 0; scar less than 2 mm/contour regularity: 1
  Suppuration Yes: 0; No: 1
  Pain VAS 6-10: 0; VAS 1-5: 1
Early healing index (remodeling phase) | at 6 weeks
  Scores are given as specified below (Hamzani et al. 2018)
  Tissue color Redder or whiter than opposite site: 0; Similar to opposite site: 1
  Scar wider than 2 mm/contour irregularity: 0; scar less than 2 mm/contour regularity: 1
  Pain VAS 6-10: 0; VAS 1-5: 1

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hamzani Y, Chaushu G. Evaluation of early wound healing scales/indexes in oral surgery: A literature review. Clin Implant Dent Relat Res. 2018 Dec;20(6):1030-1035. doi: 10.1111/cid.12680. Epub 2018 Oct 15. PMID 30324746